The prospective Nationwide Study of Perthes` Disease in Norway: Functional and Radiographic Outcomes at a Mean Follow-up of Twenty Years

# Date 01.11.2018

# Perthes study group

### Head of study group

Stefan Huhnstock
Consultant, Department for orthopaedic surgery
Oslo University Hospital
0027 Oslo

Tel. 23076017

Email: uxhuhs@ous-hf.no

### Senior investigators

Terje Terjesen
Professor emeritus dr. med
Department for orthopaedic surgery
Oslo University Hospital
0027 Oslo

Email: terje.terjesen@rikshospitalet.no

Ola Wiig PhD Department for orthopaedic surgery Oslo University Hospital 0027 Oslo

Email: olawii@ous-hf.no

The society of children's orthopaedics initiated a nationwide study on Legg- Calve Perthes disease (LCPD) in 1996. All hospitals with orthopaedic service were involved and all new diagnosed patients with LCPD were registered. Several studies (1-7) were published based on this nationwide study. Ola Wiig and Stefan Huhnstock are members of the International Perthes Study Group, Texas Scottish Rite Hospital.

### **Background**

LCPD is a juvenile hip disease which affects children between 2 and 12 years of age. It is most commonly seen boys at the age around 5-6 years. The aetiology is still unknown. The pathophysiological key event is a partial or complete disruption of the blood supply to the femoral epiphysis. The epiphyseal cartilage, the secondary ossification centre and the metaphysis undergo subsequent changes due to partial or complete osteonecrosis. In the active stages of the disease the femoral epiphysis may deform due to altered mechanical properties. At time of healing the femoral head shape may vary compared to a normal hip. Depended on the residual deformity the patients may have symptoms and complaints even after time of healing and the hip function may be impaired in young adulthood. Such a hip may also predispose for early hip osteoarthritis.

Since symptoms and hip changes are not only restricted to the active phases of the disease, it is mandatory to follow up the patients over a longer period. This study elucidates the hip function, the residual deformity and the patients reported outcome 20 years after the diagnosis with LCPD:

### Unsolved issues with LCPD

LCPD has been described for more than 100 years ago(8-10). However, there is no clear consensus on the epidemiology, aetiology the prognostic factors and treatment.

The treatment has changed dramatically in Norway over the last decades. Until the late 70s, children had been treated with traction and weight relief over several months in the active stages. Later, containment treatment was introduced and several orthotic devices had been introduced in order to maintain hip containment. Surgical Containment gained increasing popularity from the late 80s until today.

There is no consensus which treatment gives the most favourable outcomes. Several studies have been published and the results concerning the surgical (7, 11-13) or non-surgical treatment is very divergent (14-16). Most of the studies are retrospective and have a short follow up time. Those studies therefore fail to evaluate the hip shape at time of healing. The main endpoints of most of the studies are based on radiographs, leaving the functional aspect unrecognized. Thus, little is known about patient's hip function, quality of life and treatment satisfaction.

## Purpose of the study

The purpose of the study is to evaluate long term outcomes, risk factors and patient reported outcomes in young adults, 20 years after LCPD.

### Material and methods

From January 1996 until December 2000 al new diagnosed children with LCPD were registered in a nationwide Perthes study. It is a prospective, multicentre study involving 28 hospitals throughout Norway. The diagnosis was established by the local

orthopedic surgeon based on radiographic findings and clinical diagnostic. All radiographs were reviewed by Svein Svenningsen, Ola Wiig or Terje Terjesen. A total of 425 children with LCPD were involved in the study.

The study will follow up all 425 patients and it is structured in 3 phases.

# Phase 1: Follow-up of all patients in the South-Eastern Norway Regional Health Authority (HSØ)

208 patients with LCPD have been registered in HSØ(163 males) and 45 females). Average age at diagnosis was 5.8 years (1.3 - 15.2).

# Phase 2: Follow-up of all patients in the Western and Central Norway Regional Health Authorities (HVoM)

187 patients with LCPD have been registered in these two regions (141 males and 46 females). Age at diagnosis was 5.7 years (1.7 – 13.5). 93 were treated with physiotherapy, 82 were treated with surgery and 11 patients with orthosis.

# <u>Phase 3: Follow-up of all patients in the North Norway Regional Health</u> Authorities (HN)

27 patients with LCPD have been registered in this region (18 boys and 9 girls). Age at diagnosis was 6.1 years (1.8 – 13.1). 11 patients were treated with physiotherapy and 16 with orthosis.

Demographics and clinical information have been reported of all 425 patients at the initial visit. Radiographs at diagnosis, 1 year and 5 years follow-up were collected. The extent of the femoral head necrosis was evaluated with the Catterall and lateral pillar classification (17, 18). At 5 years follow-up the residual deformity was classified with the modified Stulberg's classification

The present study is planning to invite all 425 patients to a clinical and radiographic examination. The project starts in 2019 with a pilot study where 20 randomised patients will be examined.

The main study will proceed with the phases as described above. The examination will comprise a clinical visit with functional testing of the hip and radiographs of both hips.

#### Endpoints (primary /secondary)

Clinical endpoints will be the hip function and quality of life reported by the patients, using the Hip disability and Osteoarthritis Outcome Score (HOOS) (20). There will also be included functional and activity related aspects of a greater population based study in Oslo (21). Furthermore, length leg discrepancies, muscle impairment and Hip impingement tests will be performed.

<u>HOOS:</u> Validated PROM.40 questions to evaluate hip symptoms, hip function on different activity levels and quality of life.

«Oslo population study»: Scientific population study in Oslo to evaluate cardiac risks (21).

If patients would like to participate in the study, but fail to meet up for the visit, a short telephone interview will be performed including a short HOOS PS form.

#### Radiological endpoints

- a.) Stulberg classification
- b.) Coverage of the femoral head (CE angle)
- c.) Osteoarthritis Jacobsen et al.(22)
- d.) Alterations of the proximal femur (ATD, CCD)
- e.) Total hip replacement.

# **Significance**

The Norwegian Perthes study is unique in the world. It is the world largest prospective study on Perthes disease. Other long term studies on LCPD are retrospective and they do not investigate the hip function. A variety of different classifications have been used, which makes a direct comparison impossible. No study has been using PROMS in the patient assessment. The present study will be the largest prospective study on this field. It elucidates both radiographic and clinical aspects 20 years after the diagnosis. The results may therefore have a significant impact on a better understanding and the future treatment of LCPD.

### Plan

| 2018 | Identification of all pasients |
|-------------|----------------------------------------|
| 2018 - 2019 | Pilotstudy with 20 randomised pasients |
| 2019 | Dataanalysis og pilot study |
| 2019 - 2020 | Phase 1 |
| 2020 | Data analysis Phase 1 |
| 2020 – 2021 | Phase 2: |
| 2022 | Data analaysis |
| 2023 | Phase 3: |
| 2023 | Data analysis |
| 2023 - 2025 | Publication |

### Relevant literature

- 1. Wiig O, Terjesen T, Svenningsen S. Prognostic factors and outcome of treatment in Perthes' disease: a prospective study of 368 patients with five-year follow-up. J Bone Joint Surg (Br). 2008;90(10):1364-71.
- 2. Wiig O, Terjesen T, Svenningsen S. Inter-observer reliability of the Stulberg classification in the assessment of Perthes disease. Journal of children's orthopaedics. 2007;1(2):101-5.
- 3. Wiig O, Terjesen T, Svenningsen S. Inter-observer reliability of radiographic classifications and measurements in the assessment of Perthes' disease. Acta orthopaedica Scandinavica. 2002;73(5):523-30.
- 4. Huhnstock S, Svenningsen S, Pripp AH, Terjesen T, Wiig O. The acetabulum in Perthes' disease: a prospective study of 123 children. Journal of children's orthopaedics. 2014;8(6):457-65.
- 5. Huhnstock S, Svenningsen S, Pripp AH, Terjesen T, Wiig O. The acetabulum in Perthes' disease: inter-observer agreement and reliability of radiographic measurements. Acta orthopaedica. 2014;85(5):506-12.
- 6. Terjesen T, Wiig O, Svenningsen S. The natural history of Perthes' disease. Acta orthopaedica. 2010;81(6):708-14.
- 7. Terjesen T, Wiig O, Svenningsen S. Varus femoral osteotomy improves sphericity of the femoral head in older children with severe form of Legg-Calve-Perthes disease. Clin Orthop Relat Res. 2012;470(9):2394-401.
- 8. Calvé J. Sur une forme particulière de pseudo-coxalgie greffe sur des déformations caractérestiques del'extrémite supérieure du femur. Rev Chir (Paris). 1910;42:54-84.
- 9. Legg AT. An obscure affection of the hip joint. Boston Med Surg J. 1910;162:202.
- 10. Perthes GC. Über arthritis deformans juvenilis. Deutsch Z Chir 1910;107:111-59.
- 11. Wiig O, Terjesen T, Svenningsen S. Prognostic factors and outcome of treatment in Perthes' disease: a prospective study of 368 patients with five-year follow-up. The Journal of bone and joint surgery British volume. 2008;90(10):1364-71.

- 12. Herring JA, Kim HT, Browne R. Legg-Calve-Perthes disease. Part II: Prospective multicenter study of the effect of treatment on outcome. The Journal of bone and joint surgery American volume. 2004;86-A(10):2121-34.
- 13. Catterall A. The place of femoral osteotomy in the management of Legg-Calve-Perthes disease. The Hip. 1985:24-7.
- 14. Citlak A, Kerimoglu S, Baki C, Aydin H. Comparison between conservative and surgical treatment in Perthes disease. Archives of orthopaedic and trauma surgery. 2012;132(1):87-92.
- 15. Radlo W, Sulko J, Kotulski D. Outcome after conservative treatment of Perthes' disease in children. Ortopedia, traumatologia, rehabilitacja. 2004;6(5):589-94.
- 16. Rich MM, Schoenecker PL. Management of Legg-Calve-Perthes disease using an Aframe orthosis and hip range of motion: a 25-year experience. J Pediatr Orthop. 2013;33(2):112-9.
- 17. Catterall A. The natural history of Perthes' disease. The Journal of bone and joint surgery British volume. 1971;53(1):37-53.
- 18. Herring JA, Neustadt JB, Williams JJ, Early JS, Browne RH. The lateral pillar classification of Legg-Calve-Perthes disease. Journal of pediatric orthopedics. 1992;12(2):143-50.
- 19. Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. The Journal of bone and joint surgery American volume. 1969;51(4):737-55.
- 20. Klassbo M, Larsson E, Mannevik E. Hip disability and osteoarthritis outcome score. An extension of the Western Ontario and McMaster Universities Osteoarthritis Index. Scandinavian journal of rheumatology. 2003;32(1):46-51.
- 21. Holme I, Sogaard AJ, Lund-Larsen PG, Tonstad S, Haheim LL. Lonner det seg a leve sunt? Tidsskr Nor Laegeforen. 2006;126(17):2246-9.
- 22. Jacobsen S, Sonne-Holm S. Hip dysplasia: a significant risk factor for the development of hip osteoarthritis. A cross-sectional survey. Rheumatology. 2005;44(2):211-8.